CLINICAL TRIAL: NCT03821870
Title: Predictive Value of In-vitro Anti-cancer Therapy Sensitivity Testing on Tumoroids From Patients With Metastatic Pancreatic Cancer
Brief Title: Predictive Value of Analysing Tissue From Patients With Metastatic Pancreatic Cancer for Drug Sensitivity
Acronym: TIP
Status: Completed | Type: Observational
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TIP
Record Dates: First submitted 2019-01-09; First posted 2019-01-30 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Drugs, Investigational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Liver biopsy and blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Standard treatment: Standard first line treatment
  Interventions: Diagnostic Test: Inditreat; Drug: Experimental drug

INTERVENTIONS:
Diagnostic Test: Inditreat — Tumoroid formation and drug sensitivity analysis
Drug: Experimental drug — Second line treatment based on drug sensitivity analysis

SUMMARY:
It will be investigated whether it is possible to predict the effect or lack of effect of first-line treatment by analysing cancer cells from the individual patient receiving standard first line treatment. Also, the feasibility of selecting second-line therapy based on pre-treatment biopsies will be investigated.

Cells from pancreatic cancer will be grown in the laboratory to form small, circulating tumors and adjacent tissue, so called tumoroids. The tumoroids will then be exposed to different pre-specified anticancer drugs to hopefully reveal sensitivity or lack of sensitivity in the specific patient.

ELIGIBILITY:
Inclusion Criteria:

* Non-resectable pancreatic cancer

  * Biopsy proven adenocarcinoma compatible with pancreatic origin (primary tumor or metastasis)
  * If only biopsy from metastasis can be obtained, the patient must have a previously resected or image proven tumor of the pancreas
  * Deemed non-resectable at a multidisciplinary conference
* Candidate to standard systemic therapy, defined as one of

  * Gemcitabine monotherapy,
  * Gemcitabine and nab-paclitaxel combination,
  * Gemcitabine and capecitabine combination,
  * 5-fluorouracil, oxaliplatin and irinotecan combination (FOLFIRINOX), or
  * New standard treatments approved by the multidisciplinary cancer group 'Danish Pancreatic Cancer Group' in the inclusion period.
* Measurable disease according to RECIST 1.1
* ECOG performance status 0-2
* Age at least 18 years
* Adequate bone marrow, liver and renal function allowing systemic chemotherapy

  * Absolute neutrophil count ≥1.5x10^9/l and thrombocytes ≥ 100x10^9/l
  * Bilirubin ≤ 3 x upper normal value and alanine aminotransferase ≤ 5 x upper normal value
  * Calculated or measured renal glomerular filtration rate at least 30 mL/min
* Contraception for fertile women and for male patients with a fertile partner. Intrauterine device, vasectomy of a female subject's male partner or hormonal contraceptive are acceptable
* Written and orally informed consent

Exclusion Criteria:

* Potentially resectable disease

  * Incapacity, frailty, disability, or comorbidity to a degree that according to the investigator is not compatible with participation in the protocol
  * Other active malignant disease requiring therapy
  * Other systemic anti-cancer therapy (palliative radiotherapy is allowed)
  * Pregnant (positive pregnancy test) or breast feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic pancreatic cancer eligible for chemotherapy
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-02-22 (Actual)

PRIMARY OUTCOMES:
Predictive value of in-vitro testing | 2 months
  Predictive value is defined as the ability to correctly predict response or resistance to first-line chemotherapy

SECONDARY OUTCOMES:
Feasibility of selecting second-line therapy based on pre-treatment biopsies as measured by treatment response (RESIST 1.1 criteria) | Every 2 months during treatment up to 180 days
Feasibility of selecting second-line therapy based on pre-treatment biopsies as measured by progression free survival (PFS) | Every 2 months up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Lars Henrik Jensen, MD, PhD, Study Chair — Vejle Hospital
Locations (1):
- Departmen of Oncology, Vejle Hospital, Vejle, Denmark

IPD SHARING:
Plan to Share IPD: No